CLINICAL TRIAL: NCT04673383
Title: A Double-blind, Randomised, Placebo-controlled Study of Intravenous Doses of SPL026 (DMT Fumarate), a Serotonergic Psychedelic, in Healthy Subjects (Part A) and Patients With Major Depressive Disorder (Part B)
Brief Title: SPL026 (DMT Fumarate) in Healthy Subjects and MDD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Small Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT026_001
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy volunteers (active) (Experimental): SPL026 to be administered by IV injection
  Interventions: Drug: SPL026
- Healthy volunteers (placebo) (Experimental): SPL026-matched placebo to be administered by IV injection
  Interventions: Drug: Placebo
- Patients (active) (Experimental): SPL026 to be administered by IV injection
  Interventions: Drug: SPL026
- Patients (placebo) (Experimental): SPL026-matched placebo to be administered by IV injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPL026 — Intravenous solution
  Other Names: DMT; dimethyltryptamine; n,n-dimethytryptaimine
  Arms: Healthy volunteers (active); Patients (active)
Drug: Placebo — SPL026-matched placebo
  Other Names: Dummy; SPL026-matched placebo
  Arms: Healthy volunteers (placebo); Patients (placebo)

SUMMARY:
SPL026 (N,N-dimethyltryptamine [DMT] fumarate) is a psychedelic tryptamine being developed as a therapy for patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
2-part study. Part A in psychedelic-naïve healthy volunteers. Part B in patients with MDD who score moderate-severe on Ham-D.

Healthy volunteers will receive a single dose of SPL026 in a dose-escalation parallel group study.

Patients will receive up to 2 single doses of SPL026, 2 weeks apart. Dose 1 will be randomised double-blind with placebo. Dose 2 will be open label, active SPL026.

SPL026 will be administered by IV injection. Safety and tolerability, PK, PD and efficacy will be measured.

ELIGIBILITY:
Inclusion Criteria:

Normotensive male or female, deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, laboratory tests of blood and urine, Mini-International Neuropsychiatric Interview (MINI) and Beck Scale for Suicidal Ideation (BSS); willing to follow the contraception requirements of the trial; willing to refrain from psychedelic drug use (excluding the study drug) during the trial and ≥ 3 months afterwards; willing to be contacted by email and video call, and have online access; able to give fully informed written consent. Part A only: psychedelic-naïve, ie have never taken a serotonergic psychedelic drug, in any form. Must be 25 years or older. Part B only: MDD diagnosis (as per DSM-V); not on antidepressant medication or willing to discontinue antidepressant medication (eg selective serotonin reuptake inhibitor [SSRI] treatment) for a sufficient time before and during the study; no psychedelic drug use in the 6 months before dosing.

Exclusion Criteria:

Pre-menopausal females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception; clinically relevant abnormal findings at the screening assessment; acute or chronic illness (other than MDD [Part B only]) or infection; clinically relevant abnormal medical history or concurrent medical condition (other than MDD [Part B only]); positive tests for hepatitis B & C, or HIV; severe adverse reaction to any drug; use of over-the-counter or prescribed medication (excluding oral contraceptives) within previous 28 days (paracetamol [acetaminophen] permitted up to 7 days, and antidepressant medication must have ceased for at least 14 days; 28 days for MOAIs) before first dose of trial medication; drug or alcohol abuse; use of cannabis in the 24 h before each study visit; heavy smokers (> 10 [Part A] or > 20 cigarettes [Part B] daily); supine blood pressure, heart rate, or QTcF outside the acceptable ranges; participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the previous 3 months; phobia of needles or blood; possibility that volunteer will not cooperate with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in healthy volunteers | Up to three months after a single dose
  Safety and tolerability measured by lab biochemistry, adverse events and intensity rating scale to measure tolerability of the psychedelic experience
Efficacy of SPL026 in MDD patients with moderate to severe depression | 2 weeks after a single dose
  Montgomery-Åsberg Depression Rating Scale (MADRS) score (where 7 - 19 is mild depression, 20 - 34 is moderate depression, and >34 is severe depression) change from baseline at 2 weeks after the first dose (± 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: David Erritzoe, MD, Principal Investigator — Imperial College London; Malcolm Boyce, MD, Principal Investigator — Hammersmith Medicines Research; Fabian Devlin, MD, Principal Investigator — MAC Clinical Research
Locations (2):
- United Kingdom (2):
  - MAC Clinical Research, Liverpool
  - Hammersmith Medicines Research, London

IPD SHARING:
Plan to Share IPD: No
No plan for this yet.

REFERENCES:
- [Result] Good M, Joel Z, Benway T, Routledge C, Timmermann C, Erritzoe D, Weaver R, Allen G, Hughes C, Topping H, Bowman A, James E. Pharmacokinetics of N,N-dimethyltryptamine in Humans. Eur J Drug Metab Pharmacokinet. 2023 May;48(3):311-327. doi: 10.1007/s13318-023-00822-y. Epub 2023 Apr 22. PMID 37086340
- [Result] James E, Erritzoe D, Benway T, Joel Z, Timmermann C, Good M, Agnorelli C, Weiss BM, Barba T, Campbell G, Baker Jones M, Hughes C, Topping H, Boyce M, Routledge C. Safety, tolerability, pharmacodynamic and wellbeing effects of SPL026 (dimethyltryptamine fumarate) in healthy participants: a randomized, placebo-controlled phase 1 trial. Front Psychiatry. 2024 Jan 11;14:1305796. doi: 10.3389/fpsyt.2023.1305796. eCollection 2023. PMID 38274414
- See also: Clinical Trial Report Synopsis Available Here — https://www.isrctn.com/ISRCTN63465876